CLINICAL TRIAL: NCT03619837
Title: PRO-ACT: Prevention of De Novo HCV With Antiviral HCV Therapy Post-Liver
Brief Title: Prevention of De Novo HCV With Antiviral HCV Therapy Post-Liver and Post-Kidney Transplant
Acronym: PRO-ACT:
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18-24323
Record Dates: First submitted 2018-07-13; First posted 2018-08-08 (Actual); Results first posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Hepatitis C; Transplantation Disease Transmission
MeSH Terms: conditions — Hepatitis C | interventions — sofosbuvir-velpatasvir drug combination; sofosbuvir velpatasvir voxilaprevir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Arm (Experimental): Single Arm: Sofosbuvir/Velpatasvir
  Dosage: 400mg/100mg. Once daily for 12 weeks.
  Interventions: Drug: Sofosbuvir/Velpatasvir; Drug: Sofosbuvir/Velpatasvir/Voxilaprevir

INTERVENTIONS:
Drug: Sofosbuvir/Velpatasvir — Sofosbuvir/Velpatasvir starting early post-transplant for total of 12 weeks.
Drug: Sofosbuvir/Velpatasvir/Voxilaprevir — Only for patients who fail initial treatment with Sofosbuvir/Velpatasvir.
  Dosage: 400mg/100mg/100mg daily for 12 weeks.

SUMMARY:
In this study, subjects that do not have Hepatitis C virus (HCV) will be transplanted with livers or kidneys from donors who do have HCV. Medications that are used to treat HCV will be given to the study subjects shortly after transplant to protect them from developing the problems HCV can cause to the liver.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 year-old), wait-listed for primary kidney or liver transplant without a potential suitable living donor or for simultaneous liver kidney transplant;
* HCV non-infected at the time of transplant. Subjects who were previously HCV infected but who have had documented SVR12 are eligible to participate;
* Agree to use two methods of birth control during the study;
* Donor characteristics: serum HCV NAT-positive and negative for hepatitis B surface antigen. For liver transplant: pre-donation liver biopsy with no fibrosis (F0) or minimal fibrosis (F1). For kidney transplant: kidney donor profile index < 85%.

Exclusion Criteria:

* Donor and/or recipient HIV infection
* Subject pregnant or nursing
* Donor and/or recipient Hepatitis B surface antigen positive
* Kidney-pancreas transplant
* Single organ liver recipients who received hemodialysis for more than 7 days prior to liver transplantation
* Kidney recipients: on dialysis for > 5 years at time of Screening; subjects sensitized with panel reactive antibody > 80%; for single organ kidney transplant, subjects with advanced liver fibrosis (Knodell stage 3) or cirrhosis
* Individuals being treated with and needing to continue rifabutin, rifampin, carbamazepine, phenytoin, phenobarbital, oxcarbazepine, St. John's wort (Hypericum perforatum), medium- or high-dose rosuvastatin or atorvastatin, or high-dose proton pump inhibitors (See Concomitant Medications).
* Individuals treated with amiodarone within 42 days of organ transplant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2019-12-21 (Actual); Study Completion 2020-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claus Niemann, MD, Principal Investigator — University of California, San Francisco
Locations (6):
- United States (6):
  - University of California, San Francisco, San Francisco, California
  - University of Colorado Denver, Aurora, Colorado
  - Piedmont Research Institute, Atlanta, Georgia
  - Columbia University, New York, New York
  - Baylor University Medical Center - Dallas, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From July 13, 2018, to December 21, 2019, 122 patients were recruited from 6 U.S. transplant centers and completed the first part of the informed consent and were enrolled in this trial, and 24 (20%) of these received organs from HCV-viremic donors completed the second consent to receive transplant: 13 liver transplants and 11 kidney transplants.
Groups:
- Treatment Arm: Single Arm: Sofosbuvir/Velpatasvir
  Dosage: 400mg/100mg. Once daily for 12 weeks.
  Sofosbuvir/Velpatasvir: Sofosbuvir/Velpatasvir starting early post-transplant for total of 12 weeks.
  Sofosbuvir/Velpatasvir/Voxilaprevir: Only for patients who fail initial treatment with Sofosbuvir/Velpatasvir.
  Dosage: 400mg/100mg/100mg daily for 12 weeks.
Period: Screening
Arm/Group | Treatment Arm
Started | 122
Completed | 24
Not Completed | 98
Not completed — received organs from HCV-negative donors | 47
Not completed — died on the wait-list | 2
Not completed — remained on the wait list | 40
Not completed — didn't meet eligibility criteria | 3
Not completed — withdrew consent | 2
Not completed — never listed for HCV-viremic donor | 1
Not completed — developed exclusion criteria | 2
Not completed — excluded by the investigator due to non-compliance | 1
Period: Main Study
Arm/Group | Treatment Arm
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Subjects that do not have Hepatitis C virus (HCV) will be transplanted with livers or kidneys from donors who do have HCV.
Groups:
- Transplant Recipients: Single Arm: Sofosbuvir/Velpatasvir Dosage: 400mg/100mg. Once daily for12 weeks. Sofosbuvir/Velpatasvir:Sofosbuvir/Velpatasvir starting early post-transplant for total of 12 weeks.
  Sofosbuvir/Velpatasvir/Voxilaprevir:Only for patients who fail initial treatment with Sofosbuvir/Velpatasvir. [no patients failed initial treatment] Dosage: 400mg/100mg/100mg daily for12 weeks.
Arm/Group | Transplant Recipients
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 2
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57 [48 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 20
  Race: Black | 3
  Race: Asian | 1
Region of Enrollment [Number; unit: participants]
  United States | 24
Etiology of end-stage disease [Count of Participants; unit: Participants]
  nonalcohol steatohepatitis | 5
  alcohol | 4
  HCV/alcohol | 2
  alpha-1-anti-trypsin deficiency | 1
  hemochromatosis | 1
  hypertension | 4
  diabetes | 1
  polycystic disease | 2
  chronic nephritis | 2
  immunoglobulin A nephropathy | 2

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With HCV RNA Level Below Limits of Quantification (LOQ)
Description: The primary outcome was sustained virologic response, defined as HCV RNA below the lower limit of quantification 12 weeks after treatment completion (SVR12). Secondary outcomes included the proportion of patients with SVR24 defined as HCV RNA < lower limit of quantification 24 weeks after the end of treatment; with viral relapse defined as HCV RNA <LLOQ at end of treatment with subsequent quantifiable HCV RNA; and with on-treatment virologic breakthrough defined as > 1 log increase in viral RNA after treatment week 1.
  Safety was measured as the adverse events and serious adverse events attributed by the investigator to HCV infection or antiviral therapy; the proportion of recipients who prematurely discontinued antiviral therapy before the planned end of treatment; and patient and graft survival at 6 months post-transplant.
Time Frame: 12 weeks after end of treatment
Population: All patients with HC viremia documented post-transplant. 1 participant did not develop HCV viremia post transplant therefore was not included in the count of participants for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 23
Participants | 23

2. Secondary Outcome: Safety as Measured by the Proportion of Participants Who Prematurely Discontinue Antiviral Therapy Before the Planned End of Treatment
Description: 1 of 23 patients prematurely discontinued antiviral therapy due to intercurrent graft-versus-host disease that progressed to multiorgan failure.
Time Frame: 12 weeks after start of treatment
Population: 1 participant did not develop HCV viremia post transplant therefore was not included in the count of participants for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 23
Participants | 1

3. Other Pre Specified Outcome: Survival Rate of Patients and Their Allografts 6 Months Post Transplant
Description: Graft and patient survival at 24 weeks after transplant
Time Frame: 6 months from time of liver transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 24
Participants | 23

ADVERSE EVENTS:
Time Frame: 6 months
Description: AEs were graded using the Common Terminology Criteria for Adverse Events, Version 4.03, published June 2010
Groups:
- Transplant Recipients: Treatment Arm Single Arm: Sofosbuvir/Velpatasvir
  Dosage: 400mg/100mg. Once daily for 12 weeks.
Arm/Group | Transplant Recipients
All-Cause Mortality (participants affected / at risk) | 1/24
Serious Adverse Events (participants affected / at risk) | 13/24
Other Adverse Events (participants affected / at risk) | 7/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transplant Recipients (N=24)
GVHD (Immune system disorders) | 1 (1) — Subject was diagnosed with GVHD beginning day 19 following transplant. Study drug was started 8 days post_LT but was permanently discontinued after only 7 weeks of treatment per investigator discretion due to multisystem organ complications.
Rejection (Immune system disorders) | 1 (1) — Subject received an A2→O graft and began the study drug 5 days post-transplant developed early antibody-mediated rejection that was treated with intravenous immunoglobulin G with normalization of liver biochemistries by day 36 after transplant.
Biliary sclerosis (Hepatobiliary disorders) | 1 (1) — Subject who began the study drug 6 days after surgery developed a progressive, intrahepatic biliary sclerosis starting by day 31. An ischemic etiology was excluded. No other clinical sequelae other than elevated ALKP.
cardiomyopathy (Cardiac disorders) | 1 (1) — Subject started study treatment 6 days after surgery and found to have idiopathic pericardial effusion with decreased left-ventricular ejection fraction about 1 month after transplant that resolved with pericardiocentesis.
Fever (Infections and infestations) | 5 (7) — N=5 without origin; n=1 with diarrhea and n=1 with UTI
Cholangitis (Hepatobiliary disorders) | 2 (2)
Fracture (Musculoskeletal and connective tissue disorders) | 2 (2) — N=1 hip; N=1 humerus
Delayed graft function (Renal and urinary disorders) | 1 (1) — Required hemodialysis but recovered.
Ureteral stricture (Renal and urinary disorders) | 1 (1) — Associated with acute kidney injury, treated with nephrostomy with resolution
Supraventricular tachycardia (Cardiac disorders) | 1 (1) — Intraoperative with liver transplantation; treated with amiodarone
Colitis (Gastrointestinal disorders) | 1 (1) — Secondary to C. difficle
Bleeding (Surgical and medical procedures) | 2 (2) — Intraabdominal bleeding (post-op - N=2 liver transplant recipients)
Pancreatitis (Surgical and medical procedures) | 1 (1) — Post procedural
Gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1)
hyperkalemia (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transplant Recipients (N=24)
abnormal liver tests (Hepatobiliary disorders) | 5 (5)
anemia (Blood and lymphatic system disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1) — with vomiting
hematuria (Renal and urinary disorders) | 1 (1) — post kidney biopsy
Elevated creatinine (Renal and urinary disorders) | 1 (1)
leukopenia (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-18): https://cdn.clinicaltrials.gov/large-docs/37/NCT03619837/Prot_SAP_000.pdf
  • Informed Consent Form (2018-03-19): https://cdn.clinicaltrials.gov/large-docs/37/NCT03619837/ICF_001.pdf